CLINICAL TRIAL: NCT05620199
Title: Upfront Resection of Locally Advanced NSCLC Followed by Chemoradiotherapy; Phase I Multicenter Study to Assess Treatment Feasibility and Safety
Brief Title: Upfront Resection of Locally Advanced NSCLC Followed by Chemoradiotherapy
Acronym: UPLAN-I
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Leiden University Medical Center (Other); Radboud University Medical Center (Other); University Medical Center Groningen (Other); Erasmus Medical Center (Other); Maastricht University Medical Center (Other); Zuyderland Medical Centre (Other); Maxima Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M22UPL
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2022-11

CONDITIONS: Locally Advanced Non-Small Cell Lung Cancer; Chemoradiotherapy; Cavitation Lung; Surgery; Feasibility; Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study population (Experimental): All included patients will have an upfront surgery of the primary tumor, followed by chemoradiotherapy. Resection will be done within 2-4 weeks after presentation in the multidisciplinary team meeting (MDT). After resection, restaging will take place preceding start of CRT, which should start within 4-6 weeks after resection.
  Interventions: Procedure: Upfront resection

INTERVENTIONS:
Procedure: Upfront resection — Resection of the primary tumor

SUMMARY:
For patients with irresectable locally advanced non-small cell lung cancer (NSCLC) (e.g. multilevel or bulky N2 disease or presence of N3 lymph node metastases), current guidelines recommend treatment with chemoradiotherapy (CRT) followed by immune checkpoint inhibition (ICI, durvalumab). Chances of sterilization of a large (e.g. clinically staged T3 or T4 tumor) tumor volume by CRT alone are relatively small and these tumors are associated with a high local recurrence rate. Moreover, necrosis and cavitation of these tumors puts these patients at risk of fatal bleeding and might cause infectious complications, which lead to subsequent impaired quality of life (QoL) and to interruption of, or the need for postponing, (systemic) treatment.

Upfront resection of the tumor in the lung, followed by postoperative CRT in patients who have a (potentially) resectable tumor could be a strategy to prevent complications of CRT in large volume and/or cavitating tumors with extensive mediastinal disease.

DETAILED DESCRIPTION:
Stage III non-small cell lung cancer (NSCLC) comprises a heterogeneous group of patients, with concurrent chemoradiotherapy (CRT), until recently, being considered the standard of care (SoC) treatment for fit patients. Prognosis varies depending on the size and extent of the primary tumor and the degree of lymph node involvement. The aim of treatment of stage III NSCLC is to increase both locoregional and systemic control of the disease. For resectable stage III NSCLC, resection alone is associated with poor survival because of a high local recurrence rate and the presence of distant metastatic disease during the course of the disease. Induction chemotherapy and/or radiotherapy followed by surgery has been demonstrated to improve survival in selected patients. Moreover, it has been shown that in highly selected patients with stage IIIB NSCLC, surgical resection as part of multimodality therapy might be associated with improved overall survival (OS). Since a large proportion of patients with stage III NSCLC develop distant disease relapse following CRT, there is a need to treat possible presence of micrometastases and improve systemic control of the disease. Recently, immune checkpoint inhibition (ICI, durvalumab) has been added to CRT successfully and is now SoC treatment in irresectable (e.g. multilevel or bulky N2 disease or presence of N3 lymph node metastases) stage III NSCLC, leaving the role of surgery in this new treatment strategy unclear.

In large volume NSCLC and in cavitating tumors, chances of sterilization of the tumor by CRT alone are reduced, increasing the local recurrence rate, when compared to small size tumors. Between 10-20% of all lung carcinomas present with radiological cavitation, which is believed to be due to tumor necrosis as a consequence of ischemia and/or bronchial obstruction. Necrosis and cavitation of the tumor can cause infectious complications in the short and long term with subsequent impaired quality of life (QoL) and may also lead to interruption of, or the need for postponing, (systemic) treatment. Moreover, cavitation is associated with bleeding complications and even fatal pulmonary hemorrhage after CRT. Besides, lung function might be seriously impaired after CRT for a large tumor, especially in case of a centrally located tumor. It has been suggested that upfront resection with postoperative CRT in patients who have a potentially resectable tumor could be a strategy to prevent complications of tumor cavitation (e.g. infectious complications, bleeding) in large volume tumors. Moreover, in advanced NSCLC, it is suggested that (chemo)immunotherapy (or targeted therapy in case of presence of a driver mutation) improves systemic disease control, making local control of the disease more important during follow-up. To decrease the risk of a local recurrence in a situation of controlled systemic disease, local control by upfront resection of the large volume tumor might be considered.

For stage III NSCLC, immunotherapy can be added prior (neoadjuvant) or following (adjuvant) CRT. In the neoadjuvant setting, several studies have been done or are ongoing, including ICI (single agent or a combination of 2 agents) or ICI in combination with chemotherapy, radiotherapy or CRT followed by resection as a possible treatment for stage III NSCLC (NADIM(-II) trial, LCMC3 trial, NEOSTAR trial, KEYNOTE-671 trial, IMpower-030 trial, CheckMate-816, 77T trial, AEGEAN). So far, most of these studies included only a small number of patients and endpoints have been major pathological response (MPR) (<10% vital tumor present) and complete pathological response (pCR), both being surrogate markers for progression free survival (PFS) and OS. The added toxicity of ICI, especially in combination with chemotherapy, radiotherapy or CRT, still needs to be elucidated and in case of a large volume or cavitating tumor, toxicity might be related to infection and necrosis of the large tumor mass and/or an increase in radiation dose to the organs at risk such as the lungs.

Upfront surgery might benefit patients with large volume stage IIIB/IIIC NSCLC and the potential advantages, e.g. improved local control, reduction of radiotherapy treatment volumes and reduction of long term infectious problems or bleeding complications because of necrosis of the primary tumor, may possibly outweigh the risk of a delayed start of the SoC treatment. A possible drawback of an upfront resection approach is the risk of (locoregional or systemic) tumor progression when delaying planned CRT and adjuvant ICI. The intervention should not prevent the patient from receiving the SoC treatment, so a safety and feasibility check is necessary in evaluating the role of upfront resection in these patients with large volume stage IIIB/IIIC NSCLC.

Aim of the UPLAN-I trial is to evaluate feasibility and safety of upfront resection of the large volume or cavitating tumor in the lung (including hilar with/without mediastinal lymph node dissection if deemed possible by the treating surgeon), followed by concurrent CRT. The role of upfront resection in reducing infectious problems (and bleeding complications) and subsequent impaired QoL, in combination with decreasing the risk of a local recurrence (PFS) and improving OS, are evaluated in the future UPLAN-II trial, however feasibility and safety of this treatment regimen need to be established first (UPLAN-I). Moreover, the role of ctDNA in relation to treatment response and outcome of this treatment regimen will be evaluated in the consecutive UPLAN-II trial.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written and dated IC prior to any study specific procedures.
* Male or female aged at least 18 years.
* Eastern Cooperative Oncology Group (ECOG)/WHO performance status of 0 or 1.
* A pretreatment PET/CT scan (of the thorax and upper abdomen) and an MRI (or CT scan) of the brain is considered SoC and must be done prior to start of treatment.
* Pathologically proven NSCLC, staged according to the 8th edition of the AJCC Staging Manual, with a clinical indication for concurrent CRT (according to current guidelines).
* Pathology proven N2 or N3 lymph node metastasis.
* Patients should be able to receive concurrent CRT.
* Patients should be operable to the discretion of the treating pulmonary physician, surgeon and anesthesiologist, based on lung function testing and performance scoring.
* EGFR/ALK mutations and never-smokers may be included in the study (since endpoints are settled after finishing CRT and before starting adjuvant systemic treatment).

Exclusion Criteria:

* Irresectable primary lung tumor before start of concurrent CRT.
* Pneumonectomy deemed necessary (by the treating surgeon) to achieve a complete resection (R0).
* Sulcus superior tumor with invasion of the thoracic wall.
* cT3-4 based on satellite nodus/lesion in the ipsilateral lung.
* Patients with a locoregional recurrence or a second primary lung cancer.
* Patients with prior treatment with radiotherapy on the lung.
* Patients with a history of other malignancies, except:

  * adequately treated non-melanoma skin cancer
  * curatively treated in-situ cancer, or
  * other malignancies curatively treated with no evidence of disease for >5 years following the end of treatment and which, in the opinion of the treating physician, do not have a substantial risk of recurrence of the prior malignancy.
* Small cell lung cancer or a pulmonary carcinoid tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Intervention Feasibility | 2 years
  Assessed by the number of patients completing the predefined treatment. Feasibility is proven if at least 15 out of 20 patients complete the treatment protocol consisting of upfront resection and chemoradiotherapy.

SECONDARY OUTCOMES:
Intervention Safety | 2 years
  Assessed throughout the study according to CTCAE v5.0
Complications | 2 years
  Registered according to the standardized Clavien-Dindo classification of surgical complications

CONTACTS AND LOCATIONS:
Overall Officials: Koen Hartemink, MD, PhD, Principal Investigator — The Neterlands Cancer Institute (NKI), Antoni van Leeuwenhoek

IPD SHARING:
Plan to Share IPD: No
Patient data will be entered in the online electronic Case Report Form (eCRF) in a cloud-based clinical data management platform (Castor). Participant data will be encoded.